CLINICAL TRIAL: NCT02361411
Title: A Research of the Methods of Etiological Diagnosis of Cerebral Amyloid Angiopathy
Brief Title: Methods of Etiological Diagnosis of Cerebral Amyloid Angiopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Fan Dongsheng, Chairman of the department of neurolog of Peking University Third Hospital, Peking University Third Hospital
Other Study IDs: PUTH-2014191
Record Dates: First submitted 2015-02-03; First posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Cerebral Amyloid Angiopathy; Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood brain tissure
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to

1. Early identify patients based on clinical manifestation, imaging, gene and histology, explore diagnostic tools
2. get gene repertoire of Chinese
3. Build a cerebral amyloid angiopathy (CAA) prospective cohorts, observing the disease history, and exploring prognostic factors of hemorrhage in CAA patients

DETAILED DESCRIPTION:
We recruited consecutive patients with intracerebral hemorrhage(ICH). Clinical data and the results of laboratory tests and CT will be assessed and recorded. All the subjects will get gene tests including many genes related with Aβ and small vessel disease (Next-generation sequencing and target enrichment system) .

The result of the MRI Scans including cerebral microbleeds(CMBs)、Cortical superficial siderosis（cSS）, white matter change(WMC) and enlarged perivascular spaces (EPVS) will be assessed using scales. Ocular fundus exams such as funduscopy and imaging will be used to assess multiple dot and blot hemorrhages and microaneurysms by ophthalmologist. Mini-mental state examination(MMSE) will be used to assess the cognitive function.

Patients who need operation on the hematoma for the treatment will accept a brain tissue pathological exams According to this, a prospective cohort of CAA patients based on clinical manifestation, imaging, gene and histology will be built, and diagnostic tools such as gene and MRI results, etc will be explored. And we will get gene repertoire of Chinese patient with ICH.

Then, the subjects will be followed up on 30-day, 3-month, 6-month, and 1-year.The patients' clinical outcome will be assessed , and the results of laboratory tests and therapy will be recorded. Prognostic factors of patients with CAA related ICH will be explored.

ELIGIBILITY:
Inclusion Criteria:

①diagnosed wiht spontaneous cerebral hemorrhage after the head CT.

② the patients and their family members agreed to participate in this study.

Exclusion Criteria:

①cerebral hemorrhage caused by traumatic, cerebral infarction, tumor and arteriovenous malformation.

②patients who can not provide reliable information or are considered unsuitable for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We recruited consecutive patients with intracerebral hemorrhage.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
apolipoprotein E gene polymorphism | baseline

SECONDARY OUTCOMES:
CMBs were evaluated using the Microbleed Anatomical Rating Scale (MARS) | baseline
a composite outcome including multiple dot and blot hemorrhages and microaneurysms of the fundus | baseline
recurrence of cerebral hemorrhage | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China